CLINICAL TRIAL: NCT00671736
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-finding Study to Evaluate the Efficacy and Safety of Aerosolized Moli1901 in Adolescents (12 Years of Age or Older) and Adults With Cystic Fibrosis
Brief Title: Lancovutide (Moli1901) Inhalation Solution Study in Adolescents and Adults With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Nina Vartyan-Böhm, PhD, AOP Orphan Pharmaceuticals AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Moli1901-010B; EudraCT No 2006-006693-24
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; Moli1901; Lancovutide; 2622U90; duramycin; lung
MeSH Terms: conditions — Cystic Fibrosis | interventions — Moli1901; duramycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): daily inhalation
  Interventions: Drug: Moli1901
- 2 (Experimental): inhalation every other day
  Interventions: Drug: Moli1901
- 3 (Experimental): inhalation twice a week
  Interventions: Drug: Moli1901
- 4 (Placebo Comparator): daily inhalation
  Interventions: Drug: Moli1901 placebo

INTERVENTIONS:
Drug: Moli1901 — 2,5 ml inhalation solution, 8 weeks treatment period
  Other Names: Lancovutide, 2622U90, duramycin
  Arms: 1; 2; 3
Drug: Moli1901 placebo — 2,5 ml placebo solution, 8 weeks treatment period
  Arms: 4

SUMMARY:
This is a dose-finding study for the investigational product Lancovutide (Moli1901) in the exploratory phase IIb to establish minimum effective dose, optimal dose, and maximum safe dose. Additionally, the tolerability of Moli1901 shall be investigated.

DETAILED DESCRIPTION:
Study Moli1901-010B is a multi center, parallel group, placebo controlled, double-blind efficacy and safety evaluation of three different dosage schedules of aerosolized Moli1901 in adolescents (12 years of age or older), and adults. Study will start with a screening period (visit 1) followed by an 8 weeks double blind comparative treatment period (visit 2-7). Thereafter, subjects will be observed for additional 4 weeks without treatment (follow-up period and visit 8). Spirometry, pulse oximetry and other safety measurements will be performed up to 120 min after study medication inhalation. The study will be conducted in 30 sites in 9 European countries.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index
* Confirmed diagnosis of cystic fibrosis
* FEV1 between 50% and 85% of predicted
* Oxygen saturation level measured by pulse oximetry (SpO2) >90 % on room air

Exclusion Criteria:

* Bronchial hyperresponsiveness
* Unstable lung function
* Pulmonary disease such as pneumonia, tuberculosis, or lung cancer
* Acute upper respiratory tract infection within the last 2 weeks
* Acute lower respiratory tract infection (requiring antibiotics or hospitalization) within the last 4 weeks
* Pulmonary exacerbation within the last 4 weeks
* Changes from routine maintenance therapy within the last 4 weeks
* Scheduled changes to inhaled antibiotics regimen during the course of the study
* Receive or are planned to receive any treatment via "on-off" regimen (e.g. Tobramycin - TOBI®); last dose of any "on-off" treatment within the last 6 weeks
* Any clinically significant liver, renal, cardiac, neurological, or hematological disease
* ABPA or colonization with Burkholderia cepacia
* Poorly controlled diabetes mellitus

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The change in the percentage of the predicted FEV1 (forced expiratory volume in first second) value | at every study visit

SECONDARY OUTCOMES:
The ensemble of two subject reported clinical scores, which are physical dimensions of the self-report, disease-specific quality of life test, the cystic fibrosis questionnaire in the revised version | every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Eber, Prof Dr, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University, Graz, Austria

REFERENCES:
- [Background] Grasemann H, Stehling F, Brunar H, Widmann R, Laliberte TW, Molina L, Doring G, Ratjen F. Inhalation of Moli1901 in patients with cystic fibrosis. Chest. 2007 May;131(5):1461-6. doi: 10.1378/chest.06-2085. PMID 17494794
- [Background] Zeitlin PL, Boyle MP, Guggino WB, Molina L. A phase I trial of intranasal Moli1901 for cystic fibrosis. Chest. 2004 Jan;125(1):143-9. doi: 10.1378/chest.125.1.143. PMID 14718433
- [Background] Rickert DE, Dingley K, Ubick E, Dix KJ, Molina L. Determination of the tissue distribution and excretion by accelerator mass spectrometry of the nonadecapeptide 14C-Moli1901 in beagle dogs after intratracheal instillation. Chem Biol Interact. 2005 Jun 30;155(1-2):55-61. doi: 10.1016/j.cbi.2005.04.002. PMID 15893299
- [Background] McNulty MJ, Hutabarat RH, Findlay JW, Devereux K, Knick VC, Harvey RJ, Molina L. Pharmacokinetics and tissue distribution of the nonadecapeptide Moli1901 in rats and mice. Xenobiotica. 2003 Feb;33(2):197-210. doi: 10.1080/0049825021000022320. PMID 12623761
- [Background] Zebedin E, Koenig X, Radenkovic M, Pankevych H, Todt H, Freissmuth M, Hilber K. Effects of duramycin on cardiac voltage-gated ion channels. Naunyn Schmiedebergs Arch Pharmacol. 2008 Mar;377(1):87-100. doi: 10.1007/s00210-007-0248-5. Epub 2008 Jan 5. PMID 18176799
- [Derived] Eber E, Trawinska-Bartnicka M, Sands D, Bellon G, Mellies U, Bolbas K, Quattrucci S, Mazurek H, Widmann R, Schoergenhofer C, Jilma B, Ratjen F. Aerosolized lancovutide in adolescents (>/=12 years) and adults with cystic fibrosis - a randomized trial. J Cyst Fibros. 2021 Jan;20(1):61-67. doi: 10.1016/j.jcf.2020.08.014. Epub 2020 Sep 1. PMID 32888826
- See also: Sponsor — http://www.aoporphan.com/